CLINICAL TRIAL: NCT01094795
Title: A Nationwide Post-marketing Study on the Safety of Abatacept Treatment in Sweden Using the ARTIS Register
Brief Title: Safety Study of Abatacept in Sweden
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: IM101-125
Record Dates: First submitted 2010-03-24; First posted 2010-03-29 (Estimated); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Patients initiating abatacept
- Patients receiving other biologic disease-modifying drugs
- Patients with early rheumatoid arthritis (RA)
- Patients with prevalent RA identified by hospitalization
- General population

SUMMARY:
The primary purpose of this study is to assess incidence rates of targeted infections, malignancies and mortality among patients with rheumatoid arthritis who are treated with abatacept.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Sweden

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of Sweden
Sampling Method: Non-Probability Sample
Enrollment: 92635 (Actual)
Dates: Start 2011-03-31 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Hospitalized infection | Every 6 months throughout the study
Malignancy (total, lymphoma, lung cancer, breast cancer, colorectal cancer, prostate cancer) | Every 6 months throughout the study
Total mortality | Every 6 months throughout the study

SECONDARY OUTCOMES:
Autoimmune disorders (lupus, psoriasis, multiple sclerosis) | Every 6 months throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm